CLINICAL TRIAL: NCT05701735
Title: Patient Decision Aid for Chemotherapy or Exclusion in Cisplatin-Intolerant Patients With Locally Advanced Cervical Cancer (CECIL): Development, Validation and Clinical Testing
Brief Title: Decision Aid for Chemotherapy in Cisplatin-Intolerant Patients With Locally Advanced Cervical Cancer
Acronym: CECIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santo Tomas Hospital, Philippines (Other)
Collaborators: University of Santo Tomas - Graduate School (Unknown); University of Santo Tomas - Faculty of Medicine and Surgery (Unknown); University of Santo Tomas Hospital - Benavides Cancer Institute (Unknown); Philippine Council for Health Research & Development (Other Government); Manila Doctors Hospital (Network); Our Lady of Lourdes Hospital (Unknown)
Responsible Party: Principal Investigator, Warren Bacorro, Principal Investigator, University of Santo Tomas Hospital, Philippines
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: USTH-BCI-RO-2022-02
Record Dates: First submitted 2022-12-27; First posted 2023-01-27 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Locally Advanced Cervical Carcinoma
Keywords: Patient decision aid; Cervical cancer; Chemotherapy; Radiotherapy; Elderly; Renal failure; Decisional conflict
MeSH Terms: conditions — Uterine Cervical Neoplasms; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Phase 1: Embedded mixed-methods design Phase 2: Experimental, block-randomized two-arm trial design
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Given the nature of the intervention, true blinding could not be done on the participant, who is also the assessor. Blinding is necessary to control for participant expectation bias and participant performance bias. The provider (gynecologic oncologist) of the standard of care (standard consultation) is blinded to the subsequent assignment to either arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine care (No Intervention): Routine in-house workflow for initial and follow-up consultation, disclosure of diagnosis, and apprisal and counseling regarding treatment options
- Patient decision aid (Experimental): Routine in-house workflow for initial and follow-up consultation, disclosure of diagnosis, and apprisal and counseling regarding treatment options plus provision of a decision aid after the initial consultation
  Interventions: Behavioral: CECIL Patient Decision Aid

INTERVENTIONS:
Behavioral: CECIL Patient Decision Aid — The CECIL patient decision aid explicitly identifies the disease, the index decision, and the treatment options, describes the positive and negative features and consequences of each option, and guides the patient in examining personal values and preferences, to arrive at a quality and realistic decision.
  The decision aid will be developed and validated according to the guidelines and standards published by the International Patient Decision Aids Standards (IPDAS) Collaboration.
  Other Names: Decision Support Intervention
  Arms: Patient decision aid

SUMMARY:
The goal of this clinical trial is to investigate the utility and effectiveness of a decision aid in cisplatin-intolerant patients with locally advanced cervical cancer.

The main questions it aims to answer are:

1. What is the effectiveness of the decision aid in reducing decisional conflict?
2. What is the utility of the decision aid in preparing for decision-making?

Participants will be asked to accomplish the Decisional Conflict Scale before and after using the decision aid.

Researchers will compare patients given routine care and the decision aid with patients given routine care to see if the decision aid reduces decisional conflict.

DETAILED DESCRIPTION:
In locally advanced cervical cancer (LACC), adding chemotherapy (ChT) to radiotherapy (RT) improves survival at the cost of increased toxicity. Among patients with cisplatin contraindications, compliance to RT may be compromised. Shared decision-making (SDM) allows for more patient engagement in the decision-making process and decision implementation planning. In cancer-related decision-making, patient decision aids (PtDA) facilitate the SDM process and have increased patient knowledge and satisfaction and decreased decisional conflict and attitudinal barriers improved patient satisfaction and treatment compliance.

The CECIL study is a two-phase study to develop, validate and test the effectiveness of a PtDA for cisplatin-intolerant LACC patients faced with the decision of adding ChT to RT. Phase 1 is a mixed-methods study to develop a PtDA prototype and determine its content validity and user acceptability. Phase 2 is a block-randomized clinical trial to determine its effectiveness in reducing decisional conflict and its utility in preparing for decision-making. Adult women with biopsy-proven untreated LACC with cisplatin contraindications will be included in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Squamous, adeno- or adenosquamous histology
* International Federation of Gynaecology and Obstetrics (FIGO) Stage I-B3, II-A2, II-B to IV-A
* Contraindication to ChT, including but not limited to hydronephrosis, renal or cardiac dysfunction, frailty, or refusal
* Grade 6 level English literacy
* Informed consent

Exclusion Criteria:

* Other histologies
* Metastatic disease
* Other active cancers
* Prior cancer EXCEPT for a cancer treated curatively, in remission for ≥5 years, with low recurrence risk; adequately treated lentigo maligna or non-melanoma skin cancer without evidence of disease; or adequately treated carcinoma-in-situ without evidence of disease
* Prior pelvic radiotherapy, brachytherapy, or chemotherapy
* Pregnancy
* Cognitive impairment or psychological disturbance limiting study compliance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict | Prior to the second consultation visit (for treatment decision and implementation planning), usually within one week
  Decisional Conflict Scale (DCS) scores of ≥25 will indicate significant decisional conflict. The proportion of participants having pretest (baseline) and posttest decisional conflict scores of ≥25 for each group will be reported.

SECONDARY OUTCOMES:
Utility in preparation for decision-making | After use of the patient decision aid and prior to the second consultation visit (for treatment decision and implementation planning), usually within one week
  For the experimental group, the overall utility of the decision will be measured using the Preparation for Decision-Making Scale (PDMS). This will be reported as the averaged individual user mean scores using the PDMS and the confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bacorro, MD, Study Chair — University of Santo Tomas Hospital - Benavides Cancer Institute
Locations (3):
- Philippines (3):
  - Our Lady of Lourdes Hospital, Manila, National Capital Region
  - Manila Doctors Hospital, Manila, NCR
  - University of Santo Tomas Hospital, Manila, NCR

IPD SHARING:
Plan to Share IPD: Yes
All data generated in this study will remain confidential and will be stored securely at the University of Santo Tomas Hospital - Benavides Cancer Institute and will be made available upon request and upon approval of the study team.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Five years after study completion
Access Criteria: Data will only be made available to people directly involved with the study or requesting and approved parties who have signed a Confidentiality Agreement.

REFERENCES:
- [Result] Bacorro W, Baldivia K, Mariano J, Dancel E, Antonio L, Gonzalez G, Ortin TS, Canlas R. Patient Decision Aid for Chemotherapy or Exclusion in Cisplatin-Intolerant Patients With Locally Advanced Cervical Cancer: Development, Alpha Testing, and Peer Validation. JCO Glob Oncol. 2023 Sep;9:e2300096. doi: 10.1200/GO.23.00096. PMID 37677124